CLINICAL TRIAL: NCT05361590
Title: Impact of Regular Home Use of Lumoral Dual-light Photodynamic Therapy on Plaque Control and Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: Tampere University (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DPS-01
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis; Plaque, Dental; Plaque Induced Gingivitis
Keywords: Lumoral; Lumorinse; Plaque; Periodontitis; Plaque control
MeSH Terms: conditions — Periodontitis; Dental Plaque; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: 20 participants in the treatment (Lumoral) group and 20 participants in the control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects will be randomized into the study group and the control group by using a sealed envelope system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Subjects in the study group will use the Lumoral device once a day according to the verbal and written instructions provided to them. In addition, they will brush their teeth twice daily in their customary manner while using the provided sonic toothbrush and regular toothpaste.
  Interventions: Device: Lumoral device
- Control group (Active Comparator): Subjects in the control group will brush their teeth in their customary manner twice daily while using the provided sonic toothbrush and regular toothpaste. They will not receive any additional intervention.
  Interventions: Device: Lumoral device

INTERVENTIONS:
Device: Lumoral device — The Lumoral treatment -device is a CE-marked antibacterial home-use device for the treatment and prevention of oral diseases caused by bacteria. It is used in combination with a CE-marked mouth rinse called Lumorinse.
  Other Names: Lumorinse mouth rinse

SUMMARY:
This early-stage study is designed to determine the efficacy of the CE-approved, antibacterial, dual-light Lumoral method in periodontitis patients. Improved supragingival plaque control can help to also sustain the subgingival plaque management in the long term. In addition, the device might have a photobiomodulation effect on periodontal tissues.

DETAILED DESCRIPTION:
Dental plaque triggers changes in gingival health, which results in slight swelling and bleeding from the gingival margin and causes gingivitis. Supragingival dental biofilm control can be achieved by mechanical and chemical means. Toothbrushing is effective in reducing levels of dental plaque (van der Weijden & Slot 2015). It removes plaque from flat, accessible surfaces but is less effective at the gingival margins and in approximal areas, where the accumulation of residual plaque encourages gingivitis and deterioration of periodontal health. Effective toothbrushing is also depending on a number of factors, e.g., age, knowledge, manual dexterity and motivation. Oral hygiene instructions and patient motivation in oral hygiene practices should be an integral part of the patient management during all stages of periodontal treatment (Tonetti et al., 2015). Oral health practice of individuals affects their gingival and periodontal health.

The Lumoral is a CE-marked medical device developed to provide a potent, targeted antibacterial action on dental plaque in a home environment. The device mechanism of action is antibacterial photodynamic therapy. The device is used by swishing a mouth rinse, which has a strong adherence to dental plaque. The plaque-adhered photoactive mouth rinse can be activated by a simple to use light applicator. Preliminary results have shown a promising anti-inflammatory response in addition to plaque reduction.

This early-stage study is designed to determine the efficacy of the Lumoral method in periodontitis patients. Improved supragingival plaque control can help to also sustain the subgingival plaque management in the long term. In addition, the device might have a photobiomodulation effect on periodontal tissues.

Forty (40) patients are randomized to the Lumoral treatment group or the control group. Both groups shall receive standard oral hygiene instructions for sonic toothbrush, interdental brush, and dental floss use. All the patients shall be assessed for the clinical periodontal status including visible plaque index (VPI), bleeding on probing (BOP) and probing pocket depth (PPD). In addition, aMMP-8 mouth rinse test and microbiological analysis of gingival pockets will be performed. Digital photographs after staining will be taken. These analyses shall be performed at baseline and at 4 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Agreement to participate in the study and to sign a written consent form

Exclusion Criteria:

* Presence of any physical limitation or restriction that might restrict Lumoral use
* Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
BoP | 4 weeks
  Reduction in bleeding on probing (BoP).
  Procedure for BoP:
  * A full-mouth assessment at six sites per tooth
  * Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus
  * Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent"
  * BOP reported as the percentage (%) of sites with positive findings
  * Calculation formula: number of bleeding sites/ 6 times number of teeth

SECONDARY OUTCOMES:
Microbiological pathogens | 4 weeks
  Change in periodontal microbiological pathogens. The plaque sample will be taken from the teeth with ≥3 mm pockets with a sterile paper point. If the subject does not have any deep periodontal pockets, then a sample will be taken from shallow sites. Prior to sampling, the supragingival plaque will be removed with a curette. The paper point will be then taken to the gingival pocket with sterile tweezers. The paper pin will be allowed to stand for 10 to 20 seconds, after which it will be removed and sealed in an empty plastic sample transport tube.
  A gene amplification method (polymerase chain reaction, PCR) will be used to look for six key bacteria in periodontitis: Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Treponema denticola, Tannerella forsythia, Prevotella intermedia and Parvimonas micra.
aMMP-8 | 4 weeks
  Reduction in periodontal inflammation marker aMMP-8. An aMMP-8 marker analysis will be performed using Periosafe test (Dentognostics GmbH) according to the manufacturer's instructions.
VPI | 4 weeks
  Clinical improvement concerning visible plaque index (VPI).
  Procedure for VPI:
  * A full-mouth assessment, measured at 4 sites per tooth
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * VPI reported as the percentage (%) of sites with plaque
  * Calculation formula: number of sites with plaque/ 4 times number of teeth
PPD | 4 weeks
  Reduction in probing pocket depth (PPD).
  Procedure for PPD:
  * A full-mouth assessment, measured at six sites per tooth
  * Assessed from the base of the pocket to the gingival margin (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Tommi Pätilä, Docent, Study Director — Head of Research
Locations (1):
- Wellbeing services County Pirkanmaa, Health Services, Orthodontics and specialized dental care, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
The IPD will only be administered by the researchers that are listed in the CIP.

REFERENCES:
- See also: Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review. Laser Dent Sci 3, 147-153 (2019 — https://doi.org/10.1007/s41547-019-00056-9
- See also: Chapple ILC, Mealey BL, Van Dyke TE et al., (2018). Periodontal health and gingival diseases and conditions on an intact and a reduced periodontium: Consensus report of workgroup 1 of the 2017 World Workshop on the Classification of Periodontal and Peri- — https://scirp.org/reference/referencespapers.aspx?referenceid=2467179
- See also: Levine JI. Medications that increase photosensititivity. FDA document Dec 1990. — https://www.fda.gov/media/75892/download
- See also: Nikinmaa S, Alapulli H, Auvinen P, et al. (2020) Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. PLoS ONE 15(5): e0232775. — https://doi.org/10.1371/journal.pone.0232775
- See also: Lähteenmäki H, Pätilä T, Räisänen IT, et al. (2022). Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease - A Pilot Study — https://researchportal.helsinki.fi/en/publications/repeated-home-applied-dual-light-antibacterial-photodynamic-thera
- See also: Pereira PAB, Aho VTE, Paulin L, et al., (2017) Oral and nasal microbiota in Parkinson's disease. Parkinsonism and Related Disorders 38: 61-67. — http://dx.doi.org/10.1016/j.parkreldis.2017.02.026
- See also: Sanz M, Herrera D, Kebschull M, et al.; On behalf of the EFP Workshop Participants and Methodological Consultants. (2020) Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol., 47: 4- 60. — https://pubmed.ncbi.nlm.nih.gov/32383274/
- See also: Tonetti MS, Eickholz P, Loos BG et al., (2015). Principles in prevention of periodontal diseases: Consensus report of group 1 of the 11th European Workshop on Periodontology on effective prevention of periodontal and peri-implant diseases. Journal of — https://pubmed.ncbi.nlm.nih.gov/25639948/
- See also: Van der Weijden FA & Slot DE (2015). Efficacy of homecare regimens for mechanical plaque removal in managing gingivitis: A metareview. Journal of Clinical Periodontology, 42(Suppl 16), S77-S91 — https://pubmed.ncbi.nlm.nih.gov/25597787/
- See also: Gomes SC, Romagna R, Rossi V, Corvello PC, Melchiors-Angst PD. Supragingival treatment as an aid to reduce subgingival needs: a 450-day investigation Braz. oral res. 28 (1) (2014) — https://doi.org/10.1590/S1806-83242014.50000004